CLINICAL TRIAL: NCT00945022
Title: Evaluation of Safety and Efficacy of Using Lipsus Device for Oral Wetting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IMD Tech Ltd (Industry)
Responsible Party: Dr. Hanna Levy, IMD Tech Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WL - 01
Record Dates: First submitted 2009-07-13; First posted 2009-07-23 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2009-07

CONDITIONS: Oral Dryness; General Surgery
Keywords: General Surgery
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lipsus (Experimental)
  Interventions: Device: wetting lips following surgery using anesthesia

INTERVENTIONS:
Device: wetting lips following surgery using anesthesia — The investigator will position the Lipsus device in accordance with the instructions for use

SUMMARY:
Following waking up from surgery performed under general anesthesia, patients are suffering from discomforting oral dryness, and moreover, they are not allowed drinking for 24 hours. The current management involves the wetting of patient's lips using wet bandage. This action is dependent on the presence of a family member or a nurse, which is not always possible. Many patients describe the oral dryness as a suffering, added to the suffering anyway entailed by surgery.

The investigated Lipsus device is intended for oral wetting, relieving patient's suffering and minimizing the dependence on continuous presence next to patient's bed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for surgery under general anesthesia.
* Male/female age 18 and up.
* Subject able to comprehend and give informed consent for participation in this study
* Subject must sign the Informed Consent Form.

Exclusion Criteria:

* Subjects who have any form of suspicious lesion in treatment target area.
* Pregnant or lactating Subjects
* Subjects with any infection / abscess / bleeding / blister / crack / edema / fissure / ulcer / pain in treatment target area.
* Eczema or dermatitis in treatment target area
* Subjects on drugs or psychologically determined unsuitable for the study.
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol.
* Concurrent participation in any other clinical study
* Physician objection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-02 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The safety of using the Lipsus device for oral wetting will be established by physician's assessment/observation of adverse events (signs of pain, allergies, infection or any adverse effect). | 2 days

SECONDARY OUTCOMES:
The efficacy of using the Lipsus device for oral wetting will be established by Level of oral dryness improvement measured by VAS oral dryness questionnaire. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Yuskavitch, Dr., Principal Investigator — Shaari Zedek Medical Center, Jerusalem
Locations (1):
- Shaari Zedek Medical Center, Jerusalem, Israel